CLINICAL TRIAL: NCT00615147
Title: Accuracy of the D-Dimer Assay for the Exclusion of Pulmonary Embolism in a High Risk Oncologic Population: A Correlation With Ct Pulmonary Angiogram in the Urgent Care Setting
Brief Title: Accuracy of the D-Dimer Assay for the Exclusion of Pulmonary Embolism in a High Risk Oncologic Population
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 05-040
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Cancer; Pulmonary Embolism
Keywords: Any cancer; suspected pulmonary embolism
MeSH Terms: conditions — Neoplasms; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients to have a CT pulmonary angiogram for suspected pulmonary embolism will have a d-dimer drawn as is routinely done.
  Interventions: Procedure: CT pulmonary angiogram and d-dimer draw

INTERVENTIONS:
Procedure: CT pulmonary angiogram and d-dimer draw — A CT pulmonary angiogram and a d-dimer drawn within 24 hours.

SUMMARY:
The purpose of this study is to see if a blood test (D-dimer) is as precise as the CT scan for the detection of clots.

A pulmonary embolism is an obstruction of the blood vessels in your lungs usually due to a blood clot that travels to the lungs usually from the leg. Research has shown that the results of a specific blood test (D-dimer) can be used instead of a CT scan to diagnose clots. D-dimer is a valuable diagnostic marker in either detecting the presence of or monitoring the progress of blood clots. D-dimer assays have proven to be a beneficial diagnostic tool in the evaluation of patients with suspected pulmonary embolism (PE).

ELIGIBILITY:
Inclusion Criteria:

* All patients evaluated in the urgent care center and determined to need with CT pulmonary angiogram to rule out pulmonary embolism based on signs and symptoms such as dyspnea, pleuritic chest pain, tachycardia, and/or pulse oxygen desaturation will be included.

Exclusion Criteria:

* Inability to obtain CT pulmonary angiogram secondary to lack of IV access, contrast allergy or lack of consent.
* CT pulmonary angiogram not done with routine protocol for rule out pulmonary embolism.
* Less than 21 years of age

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients coming to MSKCC Urgent care unit
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2005-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The negative predictive value of the d-dimer assay relative to CT pulmonary angiogram will be the primary measure of accuracy used for this purpose. | conclusion of study

SECONDARY OUTCOMES:
To estimate the positive predictive value, sensitivity, and specificity of the d-dimer assay relative to CT pulmonary angiogram. | conclusion of study
To explore the association between the accuracy of the d-dimer assay and clinical symptoms indicating pulmonary embolism. | conclusion of study

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org